CLINICAL TRIAL: NCT04706663
Title: A Multi-Center Natural History Study of Precision-Based Genomics in Prostate Cancer
Brief Title: Precision-Based Genomics in Prostate Cancer
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000048; 000048-C
Record Dates: First submitted 2021-01-12; First posted 2021-01-13 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-26

CONDITIONS: Prostate Cancer
Keywords: germline variants; somatic variants; Genetic Predisposition; Molecular Genetics; Natural History
MeSH Terms: conditions — Prostatic Neoplasms; Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Subjects with histologically confirmed prostate cancer and genomic testing results
- Cohort 2: Subjects with histologically confirmed prostate cancer who deemed to be an exceptional responder with or without genomic testing results

SUMMARY:
Background:

Prostate cancer is the most common cancer and the second leading cause of death in males in the United States. Researchers want to find additional gene mutations that may increase a man s risk for prostate cancer and may affect how aggressive the disease is.

Objective:

To look at gene mutations in men with prostate cancer as well as the course of their disease to better understand how gene mutations relate to the way the cancer progresses and responds to treatment.

Eligibility:

Adult males 18 and older with prostate cancer who have at least one of the gene mutations researchers want to study and/or have been treated for their cancer and have had complete elimination of their cancer or stable disease for a long time.

Design:

Participants will be screened with a review of their medical records. Their gene test results will be reviewed, if available. They will be asked questions over the phone or in person.

Participants do not need to visit the NIH for this study. But if they visit NIH for another study, their data and test results will be collected. They may give blood and urine samples. They may give leftover tumor samples. These samples will be used to study their genes.

Participants who do not come to NIH on regular basis will be contacted every 6 months by phone or e-mail. They will be asked questions about their health. Data from their medical records will be collected.

Participants will have testosterone and prostate-specific antigen (PSA) tests.

Participants may be invited to NIH to give blood samples for research.

Participants on this study will be followed for life....

DETAILED DESCRIPTION:
Background:

* Prostate cancer is the most common cancer and the second leading cause of death in males in the United States with an estimated 191,930 new cases and 33,330 deaths in 2020.
* There has been progress in identifying established risk factors for the development of prostate cancer, including genetic predisposition. The study of the molecular genetics of prostate cancer has identified pathogenic variants, such as BRCA1 and BRCA2 (associated with hereditary breast and ovarian cancer syndrome), HOXB13 (associated with hereditary prostate cancer), and DNA mismatch repair (MMR) gene variants (MLH1, MSH2, MSH6, PMS2, and EPCAM) associated with Lynch syndrome.
* While our understanding of molecular genetics continues to grow, there remains a need to identify additional germline and somatic mutations and alterations that may increase an individual s risk to develop prostate cancer and potentially the aggressiveness of the disease. In studying the following alterations in prostate cancer, in both localized and advanced stages, potential expanded molecular findings may lead to actionable therapeutic targets and biomarker development. A better understanding of molecular genetics in a longitudinal study of subjects with prostate cancer may be helpful for the design of future treatment studies, and to develop a better understanding of the natural history of the disease

Objectives:

* To longitudinally evaluate subjects with prostate cancer with known germline and/or somatic variants in PIK3 and/or AKT, PALB2, BRIP1, RAD50, RAD51, RAD54, RB1, SPOP, Wnt/B-catenin pathway, CDK12, and MMR genes: MLH1, MSH2, MSH6, PMS2, and EPCAM to better understand the natural history of the disease.
* To longitudinally evaluate subjects with tumor mutational burden-high (TMB-H) prostate cancer (greater than or equal to 10 mutations/megabase [mut/Mb] or blood TMB (bTMB) [greater than or equal to16 mut/Mb]).

Eligibility:

* Subjects with histologically confirmed prostate cancer
* Must have known germline and/or somatic variants in PIK3 and/or AKT, PALB2, BRIP1, RAD50, RAD51, RAD54, RB1, SPOP, Wnt/B-catenin pathway, CDK12, and MMR genes: MLH1, MSH2, MSH6, PMS2, and EPCAM and/or TMB-high or be deemed an exceptional responder. NOTE: any platform for genomics testing is acceptable (research or CLIA-certified)
* Age greater than or equal to 18 years old

Design:

* This will be a long-term multi-center study to comprehensively study participants with prostate cancer.
* Participants will provide clinical information (including medical history, clinical tests, imaging studies and reports, surgical pathology reports, genetic test results).
* Since long-term follow-up of individuals with prostate cancer is a major feature of the study, local sites intend to maintain active contact with study subjects for as long as possible. Participants will be followed throughout the course of their illnesses, with particular attention to patterns of disease recurrence and progression, response to therapies and duration of responses.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Subjects with histologically confirmed prostate cancer.
* Must have known germline and/or somatic variants in PIK3 and/or AKT, PALB2, BRIP1, RAD50, RAD51, RAD54, RB1, SPOP, Wnt/B-catenin pathway, CDK12, and/or MMR genes: MLH1, MSH2, MSH6, PMS2, and EPCAM and/or TMB-high([defined as greater than or equal to 10 mutations/megabase (mut/Mb) and/or bTMB [greater than or equal to 16 mut/Mb]. NOTE: any platform for genomics testing is acceptable (research or CLIA-certified)

OR

* be deemed an exceptional responder. NOTE: an exceptional response is defined as achievement of either a) a complete response, or b) a confirmed partial response in a trial or treatment or a response of exceptionally long duration
* Age greater than or equal to 18 years old.
* Ability of subject to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

-None

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary clinical
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-09-14 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
natural history of prostate cancer with known germline and/or somatic variants | ongoing
  clinical presentation, patterns of disease progression, therapeutic response, disease recurrence and participant overall survival
natural history of TMB-H prostate cancer | ongoing
  clinical presentation, patterns of disease progression, therapeutic response, disease recurrence and participant overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Fatima H Karzai, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (11):
- United States (11):
  - University of California San Diego, La Jolla, California
  - University of California San Francisco, San Francisco, California
  - NorthShore University HealthSystem, Evanston, Illinois
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Dana Farber Cancer Institute, Boston, MA, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Weill Cornell Medicine, New York, New York
  - Oregon Health Sciences University, Portland, Oregon
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. @@@@@@ In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.@@@@@@Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. @@@@@@Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000048-C.html